CLINICAL TRIAL: NCT06192563
Title: A Prospective Observational Study of Adolescent Patients With Severe Atopic Dermatitis Despite Less Extensive Skin Lesions (Eczema Area and Severity Index Score < 16) Receiving Dupilumab
Brief Title: A Study to Observe How Adolescent Patients With Severe Atopic Dermatitis Despite Less Extensive Skin Lesions (Eczema Area and Severity Index Score < 16) Respond to Dupilumab Treatment
Acronym: AD-BEASCUITS
Status: Recruiting | Type: Observational
Sponsor: Sanofi (Industry)
Responsible Party: Sponsor
Other Study IDs: OBS18015; U1111-1290-5921 (Registry Identifier: ICTRP)
Record Dates: First submitted 2023-12-20; First posted 2024-01-05 (Actual); Last update posted 2024-04-15 (Actual); Status verified 2024-04

CONDITIONS: Dermatitis Atopic
MeSH Terms: conditions — Dermatitis, Atopic | interventions — dupilumab

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Adolescents with AD: Adolescent (aged 12 to 17 years) participants who suffer from severe AD with EASI score < 16, eligible for systemic dupilumab treatment according to Italian reimbursement criteria.
  Interventions: Drug: Dupilumab

INTERVENTIONS:
Drug: Dupilumab — Subcutaneous injection, standard of care as prescribed by treating physician (no investigational drug provided)
  Other Names: SAR231893 (REGN668), Dupixent®

SUMMARY:
In adolescents treated with dupilumab, clinical trials showed significant improvement of atopic dermatitis (AD) signs and symptoms, with a good safety profile. In these clinical trials, only patients with Eczema Area and Severity Index (EASI) score greater than or equal to (≥) 16 were enrolled, and effectiveness on sensitive/visible areas was not specifically evaluated. Further data about the effectiveness of dupilumab in adolescent participants with moderate to mild EASI score and severe itching and/or localized AD are therefore necessary to better understand the potential clinical benefits of dupilumab in these populations.

This is an Italian multicenter, 52-week observational (non-interventional) study which will collect data on the characteristics of adolescent (aged 12 to 17 years) participants who suffer from severe AD with EASI score less than (<) 16, eligible for systemic dupilumab treatment according to Italian reimbursement criteria. It will study the real-world effectiveness and safety of dupilumab in this population, the effect of dupilumab on itching (pruritus), sleep, quality of life and related outcomes, localized AD in sensitive/visible areas, and on coexisting atopic conditions in adolescent participants who receive dupilumab for AD. It will also document dupilumab treatment satisfaction and dupilumab discontinuation in the study participants.

DETAILED DESCRIPTION:
The individual observational period is planned to be up to 52 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Male or female, aged between 12 and 17 years at the baseline visit
* Patients with AD who have been prescribed dupilumab according to Agenzia Italiana del Farmaco (AIFA) reimbursement criteria and fulfilling the following criteria:

Patients with EASI<16 and

1. Children's Dermatology Life Quality Index (CDLQI) ≥ 10 or
2. Peak Pruritus Numerical Rating Scale (PP-NRS) ≥ 7 or
3. localization in visible or sensitive areas (head/neck/hands or genitals)

   * Patients able to understand and complete study-related questionnaires
   * Provided signed informed consent or parental/legally acceptable representative consent and patient assent where applicable

Exclusion Criteria:

* Prior use of dupilumab within 6 months prior the study entry
* Patients currently participating in any interventional clinical trial which modifies patient care
* Any condition that, in the opinion of the Investigator, may interfere with patient's ability to participate in the study (e.g., substance abuse)

The above information is not intended to contain all considerations relevant to a potential participation in a clinical trial.

Ages: 12 Years to 17 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Adolescent (aged 12 to 17 years) participants who suffer from severe AD with EASI score < 16, eligible for systemic dupilumab treatment according to Italian reimbursement criteria.
Sampling Method: Non-Probability Sample
Enrollment: 150 (Estimated)
Dates: Start 2023-11-30 (Actual); Primary Completion 2026-01-31 (Estimated); Study Completion 2026-01-31 (Estimated)

PRIMARY OUTCOMES:
Physician assessment: Percentage (%) change from baseline in Eczema Area and Severity Index (EASI) score at Week 4, Week 16 and Week 52 | Baseline, Weeks 4, 16 and 52
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicating greater severity of AD.
  EASI-50: ≥ 50% reduction in score from baseline; EASI-75: ≥ 75% reduction in score from baseline; EASI-90: ≥ 90% reduction in score from baseline.
Physician assessment: Percentage (%) of participants with EASI-50 at 4, 16, 52 weeks | Weeks 4, 16, 52
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicating greater severity of AD.
  EASI-50: ≥ 50% reduction in score from baseline; EASI-75: ≥ 75% reduction in score from baseline; EASI-90: ≥ 90% reduction in score from baseline.
Physician assessment: Percentage (%) of participants with EASI-75 at 4, 16, 52 weeks | Weeks 4, 16, 52
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicating greater severity of AD.
  EASI-50: ≥ 50% reduction in score from baseline; EASI-75: ≥ 75% reduction in score from baseline; EASI-90: ≥ 90% reduction in score from baseline.
Physician assessment: Percentage (%) of participants with EASI-90 at 4, 16, 52 weeks | Weeks 4, 16, 52
  EASI measures the severity & extent of AD based on 4 AD disease characteristics (erythema, thickness [induration, papulation, edema], scratching [excoriation] & lichenification). Total score ranges from 0 (minimum) to 72 (maximum), higher scores indicating greater severity of AD.
  EASI-50: ≥ 50% reduction in score from baseline; EASI-75: ≥ 75% reduction in score from baseline; EASI-90: ≥ 90% reduction in score from baseline.
Participant assessment: Change from baseline in Patient Oriented Eczema Measure (POEM) score at 4, 16, 52 weeks | Baseline, Weeks 4, 16, 52
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a scale ranging from 0 to 4 (0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, 4 = all days). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). Higher scores indicate more severe disease and poor quality of life.
Participant assessment: Percentage (%) of participants with a ≥ 6-point improvement from baseline in POEM score at 4, 16, 52 weeks | Baseline, Weeks 4, 16, 52
  The POEM is a 7-item self-assessment questionnaire that assesses disease symptoms on a scale ranging from 0 to 4 (0 = no days, 1 = 1 to 2 days, 2 = 3 to 4 days, 3 = 5 to 6 days, 4 = all days). The sum of the 7 items gives the total POEM score of 0 (absent disease) to 28 (severe disease). Higher scores indicate more severe disease and poor quality of life.
Percentage (%) of participants with adverse events | Baseline to Week 52
Participant assessment: Percentage (%) change from baseline in Peak Pruritus Numerical Rating Scale (PP-NRS) at 4, 16, 52 weeks | Baseline, Weeks 4, 16 and 52
  The PP-NRS is a single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD during the past 24 hours, with 0 = no itch and 10 = worst itch imaginable.
Participant assessment: Percentage (%) of participants with a ≥4-point improvement from baseline in PP-NRS at 4, 16, 52 weeks | Baseline, Weeks 4, 16 and 52
  The PP-NRS is a single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD during the past 24 hours, with 0 = no itch and 10 = worst itch imaginable.
Participant assessment: Percentage (%) of participants with a PP-NRS score of 0, 1 to 3, and 4 to 6 at 4, 16, 52 weeks (only patients with baseline PP-NRS ≥ 7 | Weeks 4, 16 and 52
  The PP-NRS is a single item 0-10 numeric rating scale assessing peak pruritus (itch) associated with AD during the past 24 hours, with 0 = no itch and 10 = worst itch imaginable.
Participant assessment: Percentage (%) change from baseline in Sleep Disturbance Numerical Rating Scale (SD-NRS) at 4, 16, 52 weeks | Baseline, Weeks 4, 16 and 52
  The SD-NRS is a single item 0-10 numeric rating scale assessing sleep disturbance associated with AD, with 0 being "no sleep loss related to the symptoms of atopic dermatitis" and 10 being "I did not sleep at all, due to the symptoms of atopic dermatitis".
Participant assessment: Percentage (%) change from baseline in Children's Dermatology Life Quality Index (CDLQI) at 4, 16, 52 weeks | Baseline, Weeks 4, 16 and 52
  The CDLQI is a validated questionnaire designed to measure the impact of skin disease on the Quality of Life. The higher the score, the greater the impact is on the quality of life.
Participant assessment: Percentage (%) of participants who achieve a ≥6-point reduction from baseline in CDLQI score at 4, 16, 52 weeks | Baseline, Weeks 4, 16 and 52
  The CDLQI is a validated questionnaire designed to measure the impact of skin disease on the Quality of Life. The higher the score, the greater the impact is on the quality of life.
Participant assessment: Percentage (%) of participants with CDLQI Score of 0 to 1, 2 to 6 and ˃ 6 at 4, 16, 52 weeks (only patients with CDLQI ≥ 10 at baseline) | Weeks 4, 16 and 52
  The CDLQI is a validated questionnaire designed to measure the impact of skin disease on the Quality of Life. The higher the score, the greater the impact is on the quality of life.
Participant assessment: Percentage (%) change from baseline in Hospital Anxiety and Depression Scale (HADS) at 4, 16, 52 weeks | Baseline, Weeks 4, 16 and 52
  The HADS is a 14-item patient-reported outcomes measure used to assess states of anxiety and depression over the past week. It is comprised of 7 items assessing anxiety and depression respectively. A Total score is out of 42 (21 per subscale). Higher scores indicate greater levels of anxiety and/or depression.
Participant assessment: Percentage (%) change from baseline Atopic Dermatitis Control Tool (ADCT) score at 4, 16, 52 weeks | Baseline, Weeks 4, 16 and 52
  ADCT is a six-item patient self-administered instrument designed and validated to assess atopic dermatitis (AD) control. The score ranges from 0-24 with higher scores indicating worsening disease control.
Participant assessment: Percentage (%) of participants with ADCT < 7 at 4, 16, 52 weeks | Weeks 4, 16 and 52
  ADCT is a six-item patient self-administered instrument designed and validated to assess atopic dermatitis (AD) control. The score ranges from 0-24 with higher scores indicating worsening disease control.
Participant assessment: Percentage (%) change from baseline the Dermatitis Family Impact (DFI) questionnaire at 4, 16, 52 weeks | Baseline, Weeks 4, 16 and 52
  The DFI is a 10-item disease specific questionnaire assessing the impact of having a child with AD on family Quality of Life (QoL). The DFI questions are scored on a four-point Likert scale ranging from 0 to 3, and the total DFI score ranges from 0 to 30. The time frame of reference is the past week, and a higher DFI score indicates greater impairment in family QoL as affected by AD.
Physician assessment: Percentage (%) of participants with Physician's Global Assessment (PGA) Face 0 or (/) 1, PGA Feet 0/1, PGA Hands 0/1, PGA Genitals 0/1 and at least a 2-point improvement from baseline at 4, 16, 52 weeks | Baseline, Weeks 4, 16 and 52
  The PGA score is a measure used in clinical practice and clinical trials to assess the severity of a particular disease. The PGA chosen for this study ranges from 0-5 point, and the following categories will be used: 0 = clear, 1 = almost clear, 2 = mild, 3 = moderate, 4 = severe, 5 = very severe. In this study, the Investigator will be evaluating four PGA scores, including PGA face, PGA feet, PGA hands, and PGA genitalia, in order to assess the severity of the localized lesions in AD patients at baseline and at week 4, 16 and 52.
Time to discontinuation and reasons for discontinuation | Baseline up to Week 52
Participant assessment: Mean score of Treatment Satisfaction Questionnaire for Medication (TSQM-9) score at 4, 16, 52 weeks | Weeks 4, 16, 52
  The 9-item TSQM (TSQM-9) is a questionnaire to assess treatment satisfaction, with scores ranging between 9 and 59, and lower scores indicating lower satisfaction with treatment.
Participant assessment: Percentage (%) change from baseline in Asthma Control Questionnaire (ACQ-6) at 4, 16, 52 weeks in participants with concomitant asthma | Baseline, Weeks 4, 16 and 52
  The ACQ-6 is a questionnaire that consists of six questions on a scale from 0 to 6 of symptoms. The questions are about limitations due to asthma and symptoms in the past week. A lower score corresponds with better asthma control.
Participant assessment: Percentage (%) change from baseline in Total Nasal Symptoms Score (TNSS) at 4, 16, 52 weeks in participants with concomitant chronic rhinitis | Baseline, Weeks 4, 16 and 52
  The TNSS is the sum of scores for each of nasal congestion, sneezing, nasal itching, and rhinorrhea using a four-point scale (0-3), where 0 indicates no symptoms, a score of 1 for mild symptoms that are easily tolerated, 2 for awareness of symptoms which are bothersome but tolerable and 3 is reserved for severe symptoms that are hard to tolerate and interfere with daily activity. TNSS is calculated by adding the score for each of the symptoms to a total out of 12.

CONTACTS AND LOCATIONS:
Overall Officials: Clinical Sciences & Operations, Study Director — Sanofi
Locations (9):
- Italy (9):
  - Investigational Site Number: 002, Bologna
  - Investigational Site Number: 006, Brescia
  - Investigational Site Number: 004, Florence
  - Investigational Site Number: 001, Milan
  - Investigational Site Number: 010, Napoli
  - Investigational Site Number: 011, Napoli
  - Investigational Site Number: 005, Roma
  - Investigational Site Number: 009, Roma
  - Investigational Site Number: 014, Verona

IPD SHARING:
Plan to Share IPD: Yes
Qualified researchers may request access to patient level data and related study documents including the clinical study report, study protocol with any amendments, blank case report form, statistical analysis plan, and dataset specifications. Patient level data will be anonymized and study documents will be redacted to protect the privacy of trial participants. Further details on Sanofi's data sharing criteria, eligible studies, and process for requesting access can be found at: https://vivli.org